CLINICAL TRIAL: NCT05845645
Title: A 2-Part Study to Evaluate the Relative Bioavailability of 2 New Formulations of UCB0599 and the Effect of Esomeprazole on the PK of UCB0599 in Healthy Participants (Part A, Open-Label) and to Assess the Safety/Tolerability and PK of UCB0599 in Healthy Participants of Japanese and Chinese Origins (Part B, Double-Blind)
Brief Title: A Study to Test Bioavailability of of 2 New Formulations of UCB0599 in Healthy Participants in Part A and to Test Safety, Tolerability, and Pharmacokinetic (PK) of UCB0599 in Healthy Japanese and Chinese Participants in Part B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0073
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy Study Participants
Keywords: Phase 1; Healthy Study Participants; UCB0599; Bioavailability study
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: Part A of the study is following a full crossover design and Part B is a parallel design with crossover character referring to the dose levels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A is open-label and Part B double-blind (Participants will be blinded to the treatment (ie, UCB0599 or Placebo), but not to the dosage).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Experimental): Study participants enrolled and randomized to this arm will receive a single dose of UCB0599 in 3 different formulations according to a pre-specified sequence during both Treatment Periods in the absence of esomeprazole, and the Treatment Periods in the presence of esomeprazole.
  Interventions: Drug: UCB0599; Other: Esomeprazole
- Part B (Experimental): Study participants enrolled to this arm will receive pre-specified doses of UCB0599 or Placebo in a pre-specified sequence during the Treatment Period.
  Interventions: Drug: UCB0599; Other: Placebo

INTERVENTIONS:
Drug: UCB0599 — Study participants will receive pre-specified doses of UCB0599 in 3 different formulations administered orally in a pre-specified sequence during the Treatment Periods of Part A and B
Other: Esomeprazole — Study participants will receive fixed dose of esomeprazole administered orally in a pre-specified sequence during the Treatment Period of Part A. This is a non-investigational medicinal product (NIMP) in this study.
  Arms: Part A
Other: Placebo — Study participants will receive placebo comparator administered orally in a a pre-specified sequence during the Treatment Period of Part B.
  Other Names: PBO
  Arms: Part B

SUMMARY:
The purpose of the study is to estimate the relative bioavailability of 2 new UCB0599 formulations under elevated and normal gastric pH conditions in healthy participants (Part A) and to asess the safety, tolerability and pharmacokinetics of UCB0599 in healthy participants of Japanese and Chinese origins (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Part A only: all healthy study participants except for those participants who are eligible for Part B of the study
* For participants of Japanese origin (Part B): study participant is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (a participant has all 4 Japanese grandparents born in Japan). For participants of Chinese origin (Part B): study participant is of Chinese descent as evidenced by appearance and verbal confirmation of familial heritage (a participant has all 4 Chinese grandparents born in China).
* Body weight within 45 to 100 kg (female) and 50 to 100 kg (male) and body mass index (BMI) within the range 18 to 30 kg/m^2 (inclusive at screening)
* Healthy male and female study participants

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Participant has a history or presence of/significant history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Participant has had lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell carcinomas that have been resected, squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Participant has had breast cancer within the past 10 years
* Participant has a history of alcohol or drug abuse within the last 1 year from Screening, as defined according to the Diagnostic and Statistical Manual of Mental Disorders
* Participant has a known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol
* Participant has a consumption of more than 600 mg of caffeine/day at screening and throughout the study
* Participant has consumed any grapefruit, grapefruit juice, grapefruit-containing products, or star fruit within 14 days prior to administration of study medication or is not willing to refrain from consuming these products for the duration of the study
* Participant has previously participated in this study or participant has previously been assigned to treatment in a study of the medication under investigation in this study
* Participant has participated in another study of a study medication (and/or an investigational device) within the previous 30 days or 5 half-lives, whichever is greatest, or is currently participating in another study of an study medication (and/or an investigational device)
* Presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to dosing
* Positive hepatitis C antibody test (HCVAb) result at screening or within 3 months prior to starting study intervention
* Positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study medication
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* For women of childbearing potential, study participant is pregnant, planning on becoming pregnant during the study, or is breastfeeding
* Participants who may have a history of confirmed gastric ulceration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0073 10001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in May 2023 and concluded in April 2024.
Pre-assignment Details: The Participant Flow refers to the Randomized Set Part A and Randomized Set Part B. Part A: P1, P2, P3, P4, P5, and P6 refer to period 1 to 6.
Groups:
- Part A: Treatment Sequence: ABC: Participants received a single dose of UCB0599 180 milligrams (mg) capsule (reference) (Treatment A) under fasting conditions on Day 1 in Period (P) 1 (normal gastric pH) and Day 19 in Period 4 (elevated gastric pH), followed by a single dose of UCB0599 180 mg non-encapsulated tablet (Treatment B) under fasting conditions on Day 6 in Period 2 (normal gastric pH) and Day 24 in Period 5 (elevated gastric pH), further followed by a single dose of UCB0599 180 mg encapsulated tablet (Treatment C) under fasting conditions on Day 11 in Period 3 (normal gastric pH) and Day 29 in Period 6 (elevated gastric pH). In Periods 4, 5, and 6 (elevated gastric pH), esomeprazole 40 mg was coadministered once daily from Day 14 to Day 33. Each treatment period was followed by a 4-day Washout period.
- Part A: Treatment Sequence: ACB: Participants received a single dose of UCB0599 180 mg capsule (reference) (Treatment A) under fasting conditions on Day 1 in Period 1 (normal gastric pH) and Day 19 in Period 4 (elevated gastric pH), followed by a single dose of UCB0599 180 mg encapsulated tablet (Treatment C) under fasting conditions on Day 6 in Period 2 (normal gastric pH) and Day 24 in Period 5 (elevated gastric pH), further followed by a single dose of UCB0599 180 mg non-encapsulated tablet (Treatment B) under fasting conditions on Day 11 in Period 3 (normal gastric pH) and Day 29 in Period 6 (elevated gastric pH). In Periods 4, 5, and 6 (elevated gastric pH), esomeprazole 40 mg was coadministered once daily from Day 14 to Day 33. Each treatment period was followed by a 4-day Washout period.
- Part A: Treatment Sequence: BCA: Participants received a single dose of UCB0599 180 mg non-encapsulated tablet (Treatment B) under fasting conditions on Day 1 in Period 1 (normal gastric pH) and Day 19 in Period 4 (elevated gastric pH), followed by a single dose of UCB0599 180 mg encapsulated tablet (Treatment C) under fasting conditions on Day 6 in Period 2 (normal gastric pH) and Day 24 in Period 5 (elevated gastric pH), further followed by a single dose of UCB0599 180 mg capsule (Treatment A) under fasting conditions on Day 11 in Period 3 (normal gastric pH) and Day 29 in Period 6 (elevated gastric pH). In Periods 4, 5, and 6 (elevated gastric pH), esomeprazole 40 mg was coadministered once daily from Day 14 to Day 33. Each treatment period was followed by a 4-day Washout period.
- Part A: Treatment Sequence: BAC: Participants received a single dose of UCB0599 180 mg non-encapsulated tablet (Treatment B) under fasting conditions on Day 1 in Period 1 (normal gastric pH) and Day 19 in Period 4 (elevated gastric pH), followed by a single dose of UCB0599 180 mg capsule under fasting conditions (Treatment A) on Day 6 in Period 2 (normal gastric pH) and Day 24 in Period 5 (elevated gastric pH), further followed by a single dose of UCB0599 180 mg encapsulated tablet (Treatment C) under fasting conditions on Day 11 in Period 3 (normal gastric pH) and Day 29 in Period 6 (elevated gastric pH). In Period 4,5 and 6 (elevated gastric pH) esomeprazole 40 mg once daily was coadministered from day 14 to 33. Each treatment period was followed by a 4-day Washout Period.
- Part A: Treatment Sequence: CAB: Participants received a single dose of UCB0599 180 mg encapsulated tablet (Treatment C) under fasting conditions on Day 1 in Period 1 (normal gastric pH) and Day 19 in Period 4 (elevated gastric pH), followed by a single dose of UCB0599 180 mg capsule (Treatment A) under fasting conditions on Day 6 in Period 2 (normal gastric pH) and Day 24 in Period 5 (elevated gastric pH), further followed by a single dose of UCB0599 180 mg non-encapsulated tablet (Treatment B) under fasting conditions on Day 11 in Period 3 (normal gastric pH) and Day 29 in Period 6 (elevated gastric pH). In Periods 4, 5, and 6 (elevated gastric pH), esomeprazole 40 mg was coadministered once daily from Day 14 to Day 33. Each treatment period was followed by a 4-day Washout period.
- Part A: Treatment Sequence: CBA: Participants received a single dose of UCB0599 180 mg encapsulated tablet (Treatment C) under fasting conditions on Day 1 in Period 1 (normal gastric pH) and Day 19 in Period 4 (elevated gastric pH), followed by a single dose of UCB0599 180 mg non-encapsulated tablet (Treatment B) under fasting conditions on Day 6 in Period 2 (normal gastric pH) and Day 24 in Period 5 (elevated gastric pH), further followed by a single dose of UCB0599 180 mg capsule (Treatment A) under fasting conditions on Day 11 in Period 3 (normal gastric pH) and Day 29 in Period 6 (elevated gastric pH). In Periods 4, 5, and 6 (elevated gastric pH), esomeprazole 40 mg was coadministered once daily from Day 14 to Day 33. Each treatment period was followed by a 4-day Washout period.
- Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg: Participants received a single dose of UCB0599 matching placebo 90 mg capsule on Day 1 in Period 1, followed by a single dose of UCB0599 matching placebo 180 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a washout period of 4 days.
- Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg: Participants received a single dose of UCB0599 90 mg capsule on Day 1 in Period 1 followed by a single dose of UCB0599 180 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a wash out period of 4 days.
- Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg: Participants received a single dose of UCB0599 matching placebo 180 mg capsule on Day 1 in Period 1 followed by a single dose of UCB0599 matching placebo 360 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a wash out period of 4 days.
- Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg: Participants received a single dose of UCB0599 180 mg capsule on Day 1 in Period 1 followed by a single dose of UCB0599 360 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a wash out period of 4 days.
- Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg: Participants received a single dose of UCB0599 matching placebo 360 mg capsule on Day 1 in Period 1 followed by a single dose of UCB0599 matching placebo 90 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a wash out period of 4 days.
- Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg: Participants received a single dose of UCB0599 360 mg capsule on Day 1 in Period 1 followed by a single dose of UCB0599 90 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a wash out period of 4 days.
Period: Part A: P1 (Day 1, Normal Gastric pH)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: P2 (Day 6, Normal Gastric pH)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: P3 (Day 11, Normal Gastric pH)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: P4 (Day 19,Elevated Gastric pH)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: P5 (Day 24,Elevated Gastric pH)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 7 | 7 | 7 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 6 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Consent Withdrawn (not due to adverse event) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: P6 (Day 29,Elevated Gastric pH)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 7 | 7 | 6 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 6 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B- Period 1 (Day 1)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 2 | 9 | 2 | 8
Japnese Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 4 | 1 | 4
Chinese Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 5 | 1 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 2 | 8 | 2 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part B- Period 2 (Day 6)
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Placebo 90 mg/Placebo 180 mg | Part B: Treatment Sequence: UCB0599 90 mg/UCB0599 180 mg | Part B: Treatment Sequence: Placebo 180 mg/Placebo 360 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence:Placebo 360 mg/Placebo 90 mg | Part B: Treatment Sequence: UCB0599 360 mg/ UCB0599 90 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 2 | 8 | 2 | 8
Japnese Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 4 | 1 | 4
Chinese Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 4 | 1 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 2 | 8 | 2 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Sets (Part A & B) included all study participants who were randomized and received full or partial study medication according to the treatment that the participants actually received.
Groups:
- Part B: Treatment Sequence: Pooled Placebo: Participants received UCB0599 matching placebo, 90 mg capsule, on Day 1 in Period 1 followed by UCB0599 matching placebo, 180 mg capsule, on Day 6 in Period 2; received UCB0599 matching placebo, 180 mg capsule, on Day 1 in Period 1 followed by UCB0599 matching placebo, 360 mg capsule, on Day 6 in Period 2; and UCB0599 matching placebo, 360 mg capsule, on Day 1 in Period 1 followed by UCB0599 matching placebo, 90 mg capsule, on Day 6 in Period 2. Arm sequences were pooled for placebo in Part B.
- Part B: Treatment Sequence: UCB0599 90mg/UCB0599 180 mg: received a single dose of UCB0599 90 mg capsule on Day 1 in Period 1 followed by a single dose of UCB0599 180 mg capsule on Day 6 in Period 2 under fasting conditions. Periods 1 and 2 were separated by a wash out period of 4 days.
- Part B: Treatment Sequence: UCB0599 360mg/ UCB0599 90mg: Participants received UCB0599 360 mg capsule, on Day 1 in Period 1 followed by UCB0599 90 mg capsule, on Day 6 in Period 2.
- Total: Total of all reporting groups
Arm/Group | Part A: Treatment Sequence: ABC | Part A: Treatment Sequence: ACB | Part A: Treatment Sequence: BCA | Part A: Treatment Sequence: BAC | Part A: Treatment Sequence: CAB | Part A: Treatment Sequence: CBA | Part B: Treatment Sequence: Pooled Placebo | Part B: Treatment Sequence: UCB0599 90mg/UCB0599 180 mg | Part B: Treatment Sequence: UCB0599 180 mg/ UCB0599 360 mg | Part B: Treatment Sequence: UCB0599 360mg/ UCB0599 90mg | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 6 | 8 | 9 | 8 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 7 | 7 | 7 | 7 | 6 | 8 | 9 | 8 | 73
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (7.1) | 42.6 (7.4) | 37.0 (10.9) | 30.9 (5.5) | 33.1 (8.8) | 31.9 (8.7) | 39.5 (9.8) | 39.3 (7.9) | 30.7 (6.5) | 40.1 (9.0) | 36.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 1 | 3 | 4 | 1 | 2 | 1 | 2 | 27
  Male | 3 | 1 | 4 | 6 | 4 | 3 | 5 | 6 | 8 | 6 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 9 | 8 | 31
  Black | 3 | 1 | 1 | 5 | 1 | 2 | 0 | 0 | 0 | 0 | 13
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 6 | 6 | 2 | 5 | 5 | 0 | 0 | 0 | 0 | 28
  Other or Mixed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 3 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 16
  Not Hispanic or Latino | 4 | 4 | 4 | 6 | 4 | 4 | 6 | 8 | 9 | 8 | 57

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of UCB0599 in Part A
Description: Cmax was maximum (peak) observed drug concentration following a single dose administration of UCB0599 under normal and elevated gastric pH condition.
Time Frame: Predose and at 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, and 96 hours after UCB0599 administration on Days 1, 6, 11, 19, 24 and 29 in Part A
Population: Pharmacokinetic Set Part A (PKS A) included all randomized participants who received at least 1 total dose of study medication and have at least 1 observable PK measurement. Here, "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A: UCB0599: Capsule 180 mg: All participants who received a single dose of UCB0599 180 mg capsule under fasting conditions on Day 1 in Period 1 (normal gastric pH), Day 19 in Period 4 (elevated gastric pH), Day 11 in Period 3 (normal gastric pH), Day 29 in Period 6 (elevated gastric pH), Day 6 in Period 2 (normal gastric pH), and Day 24 in Period 5 (elevated gastric pH). Esomeprazole was coadministered with UCB0599 180 mg capsule in Treatment Periods 4, 5, and 6 (elevated gastric pH).
- Part A: UCB0599: Non-encapsulated Tablet 180 mg: All participants who received a single dose of UCB0599 180 mg non-encapsulated tablet under fasting conditions on Day 1 in Period 1 (normal gastric pH), Day 19 in Period 4 (elevated gastric pH), Day 6 in Period 2 (normal gastric pH), Day 24 in Period 5 (elevated gastric pH), Day 11 in Period 3 (normal gastric pH), and Day 29 in Period 6 (elevated gastric pH). Esomeprazole was coadministered with UCB0599 180 mg non-encapsulated tablet in Treatment Periods 4, 5, and 6 (elevated gastric pH).
- Part A: UCB0599: Encapsulated Tablet 180 mg: All participants who received a single dose of UCB0599 180 mg encapsulated tablet under fasting conditions on Day 1 in Period 1 (normal gastric pH), Day 19 in Period 4 (elevated gastric pH), Day 6 in Period 2 (normal gastric pH), Day 24 in Period 5 (elevated gastric pH), Day 11 in Period 3 (normal gastric pH), and Day 29 in Period 6 (elevated gastric pH). Esomeprazole was coadministered with UCB0599 180 mg encapsulated tablet in Treatment Periods 4, 5, and 6 (elevated gastric pH).
Arm/Group | Part A: UCB0599: Capsule 180 mg | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599: Encapsulated Tablet 180 mg
Number analyzed (Participants) | 42 | 42 | 42
nanograms per milliliter (ng/mL)
  Normal | 876.2 (30.2) | 724.6 (39.4) | 618.0 (38.2)
  Elevated: number analyzed (Participants) | 41 | 40 | 42
  Elevated | 449.3 (54.9) | 694.4 (43.8) | 631.4 (42.8)
Statistical Analysis 1: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Non-encapsulated Tablet 180 mg; For normal gastric pH; Test type: Other; GLSM Ratio = 0.8269, 90% CI 2-sided [0.7535 to 0.9076] — The geometric least square mean (GLSM) ratio was calculated as UCB0599: Non-encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 2: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.7053, 90% CI 2-sided [0.6427 to 0.7741] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 3: Comparison: Part A: UCB0599: Non-encapsulated Tablet 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.8529, 90% CI 2-sided [0.7771 to 0.9361] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Non-encapsulated tablet 180 mg
Statistical Analysis 4: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Non-encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 1.563, 90% CI 2-sided [1.376 to 1.776] — The GLSM ratio was calculated as UCB0599: Non-encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 5: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 1.415, 90% CI 2-sided [1.248 to 1.604] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 6: Comparison: Part A: UCB0599: Non-encapsulated Tablet 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 0.9050, 90% CI 2-sided [0.7972 to 1.027] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Non-encapsulated tablet 180 mg

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC(0-t)) of UCB0599 in Part A
Description: AUC(0-t) was area under the plasma concentration-time curve from time 0 to the last quantifiable concentration of UCB0599 under normal and elevated gastric pH condition.
Time Frame: as for outcome 1
Population: PKS A included all randomized participants who received at least 1 total dose of study medication and have at least 1 observable PK measurement. Here, "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour nanograms per milliliter (h*ng/mL)
Arm/Group | Part A: UCB0599: Capsule 180 mg | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599: Encapsulated Tablet 180 mg
Number analyzed (Participants) | 42 | 42 | 42
hour nanograms per milliliter (h*ng/mL)
  Normal | 5774 (35.5) | 5503 (41.0) | 5324 (43.1)
  Elevated: number analyzed (Participants) | 41 | 40 | 42
  Elevated | 5489 (49.2) | 5779 (43.9) | 5641 (41.3)
Statistical Analysis 1: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Non-encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.9529, 90% CI 2-sided [0.9052 to 1.003] — The GLSM ratio was calculated as UCB0599: Non-encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 2: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.9220, 90% CI 2-sided [0.8758 to 0.9706] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 3: Comparison: Part A: UCB0599: Non-encapsulated Tablet 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.9676, 90% CI 2-sided [0.9191 to 1.019] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Non-encapsulated tablet 180 mg
Statistical Analysis 4: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Non-encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 1.059, 90% CI 2-sided [1.001 to 1.120] — The GLSM ratio was calculated as UCB0599: Non-encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 5: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 1.038, 90% CI 2-sided [0.9826 to 1.097] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 6: Comparison: Part A: UCB0599: Non-encapsulated Tablet 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 0.9804, 90% CI 2-sided [0.9273 to 1.037] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Non-encapsulated tablet 180 mg

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC Inf) of UCB0599 in Part A
Description: AUC inf was area under the plasma concentration-time curve from time 0 to infinity of UCB0599 under normal and elevated gastric pH condition.
Time Frame: as for outcome 1
Population: PKS A included all randomized participants who received at least 1 total dose of study medication and have at least 1 observable PK measurement. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: UCB0599: Capsule 180 mg | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599: Encapsulated Tablet 180 mg
Number analyzed (Participants) | 40 | 39 | 42
h*ng/mL
  Normal: number analyzed (Participants) | 39 | 39 | 40
  Normal | 5829 (36.8) | 5561 (42.3) | 5374 (44.5)
  Elevated: number analyzed (Participants) | 40 | 38 | 42
  Elevated | 5538 (49.5) | 5835 (44.9) | 5720 (41.4)
Statistical Analysis 1: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Non-encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.9519, 90% CI 2-sided [0.9011 to 1.006] — The GLSM ratio was calculated as UCB0599: Non-encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 2: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.9255, 90% CI 2-sided [0.8762 to 0.9777] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 3: Comparison: Part A: UCB0599: Non-encapsulated Tablet 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Normal gastric pH; Test type: Other; GLSM ratio = 0.9723, 90% CI 2-sided [0.9204 to 1.027] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Non-encapsulated tablet 180 mg
Statistical Analysis 4: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Non-encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 1.053, 90% CI 2-sided [0.9940 to 1.116] — The GLSM ratio was calculated as UCB0599: Non-encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 5: Comparison: Part A: UCB0599: Capsule 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 1.027, 90% CI 2-sided [0.9710 to 1.086] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Capsule 180 mg
Statistical Analysis 6: Comparison: Part A: UCB0599: Non-encapsulated Tablet 180 mg vs Part A: UCB0599: Encapsulated Tablet 180 mg; For Elevated gastric pH; Test type: Other; GLSM ratio = 0.9747, 90% CI 2-sided [0.9208 to 1.032] — The GLSM ratio was calculated as UCB0599: Encapsulated tablet 180 mg divided by UCB0599: Non-encapsulated tablet 180 mg

4. Primary Outcome: Percentage of Study Participants With Treatment-emergent Adverse Events (TEAEs) in Part B
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE was defined as AEs starting on/after the date/time of first treatment & upto including 4 days after last treatment or any unresolved event already present before administration of treatment that worsens in intensity following exposure to treatment.
Time Frame: From Baseline (Day 1) to Safety Follow-up Period of Part B (up to Day 15)
Population: Safety Set Part B (SS B) included all study participants who were randomized and received full or partial study medication according to the treatment that the participants actually received.
Measure: Number; unit: percentage of participants
Groups:
- Part B: Pooled Placebo (Japanese Participants): All the Japanese participants who received placebo (matching to UCB0599 90 mg, 180 mg, 360 mg) on Day 1 of Period 1 and Day 6 of Period 2. Pooled data is reported for the placebo group.
- Part B: UCB0599 90 mg (Japanese Participants): Japanese participants who received a single dose of UCB0599 90 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
- Part B: UCB0599 180 mg (Japanese Participants): Japanese participants who received a single dose of UCB0599 180 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
- Part B: UCB0599 360 mg (Japanese Participants): Japanese participants who received a single dose of UCB0599 360 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
- Part B: Pooled Placebo (Chinese Participants): All the Chinese participants who received placebo (matching to UCB0599 90 mg, 180 mg, 360 mg) on Day 1 of Period 1 and Day 6 of Period 2. Pooled data is reported for the placebo group.
- Part B: UCB0599 90 mg (Chinese Participants): Chinese participants received a single dose of UCB0599 90 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
- Part B: UCB0599 180 mg (Chinese Participants): Chinese participants received a single dose of UCB0599 180 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
- Part B: UCB0599 360 mg (Chinese Participants): Chinese participants received a single dose of UCB0599 360 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
Arm/Group | Part B: Pooled Placebo (Japanese Participants) | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360 mg (Japanese Participants) | Part B: Pooled Placebo (Chinese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 3 | 8 | 9 | 8
percentage of participants | 33.3 | 25.0 | 0 | 0 | 33.3 | 12.5 | 33.3 | 25.0

5. Primary Outcome: Percentage of Study Participants With Serious Treatment-emergent Adverse Events (Serious TEAEs) in Part B
Description: Serious TEAEs were any untoward medical incidence in a participant during administered study treatment, whether or not these events were related to study treatment and additionally were emergent untoward medical occurrence that at any dose:
  1. Results in death
  2. Is life-threatening
  3. Required in patient hospitalisation or prolongation of existing hospitalisation
  4. Results in persistent disability/incapacity
  5. Was a congenital anomaly or birth defect
  6. Important medical events
Time Frame: From Baseline (Day 1) to Safety Follow-up Period of Part B (up to Day 15)
Population: SS B included all study participants who were randomized and received full or partial study medication according to the treatment that the participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Pooled Placebo (Japanese Participants) | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360 mg (Japanese Participants) | Part B: Pooled Placebo (Chinese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 3 | 8 | 9 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage of Study Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From Study in Part B
Description: : An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE was defined as AEs starting on/after the date/time of first treatment & upto including 4 days after last treatment or any unresolved event already present before administration of treatment that worsens in intensity following exposure to treatment.
Time Frame: From Baseline (Day 1) to Safety Follow-up Period of Part B (up to Day 15)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Groups:
- Part B: UCB0599 180 mg (Japanese Participants); Part B: UCB0599 360 mg (Japanese Participants): Japanese participants who received a single dose of UCB0599 360 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
- Part B: UCB0599 180 mg (Chinese Participants): Chinese participants received a single dose of UCB0599 180 mg capsule Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
Arm/Group | Part B: Pooled Placebo (Japanese Participants) | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360 mg (Japanese Participants) | Part B: Pooled Placebo (Chinese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 3 | 8 | 9 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Maximum Plasma Concentration (Cmax) of UCB0599 in Part B
Description: Cmax was maximum (peak) observed drug concentration following a single dose administration of UCB0599.
Time Frame: Predose and at 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, and 96 hours after UCB0599 administration on Days 1, and 6 in Part B
Population: Pharmacokinetic Set Part B (PKS B) included randomized participants who received at least 1 total dose of study medication and have at least 1 observable PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360 mg (Japanese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 8
ng/mL | 502.5 (29.8) | 602.9 (42.4) | 1757 (36.4) | 483.2 (42.6) | 737.5 (35.7) | 1525 (24.8)

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC(0-t)) of UCB0599 in Part B
Description: AUC(0-t) was area under the plasma concentration-time curve from time 0 to the last quantifiable concentration of UCB0599.
Time Frame: as for outcome 7
Population: The PKS B included randomized participants who received at least 1 total dose of study medication and have at least 1 observable PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360 mg (Japanese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 8
h*ng/mL | 3363 (29.5) | 5242 (23.6) | 12010 (36.5) | 3795 (23.5) | 6689 (28.6) | 14020 (25.2)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC (Inf)) of UCB0599 in Part B
Description: AUC inf was area under the plasma concentration-time curve from time 0 to infinity of UCB0599.
Time Frame: as for outcome 7
Population: The PKS B included randomized participants who received at least 1 total dose of study medication and have at least 1 observable PK measurement. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360 mg (Japanese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
Number analyzed (Participants) | 8 | 6 | 8 | 8 | 9 | 8
h*ng/mL | 3425 (29.6) | 5151 (27.5) | 12100 (36.7) | 3847 (23.2) | 6741 (28.5) | 14070 (25.1)

10. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Adverse Events (TEAEs) in Part A
Description: as for outcome 4
Time Frame: From Baseline (Day 1) to Safety Follow-up Period of Part A (up to Day 39)
Population: Safety Set Part A (SS A) included all study participants who were randomized and received full or partial study medication according to the treatment that the participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: UCB0599: Capsule 180 mg | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599: Encapsulated Tablet 180 mg
Number analyzed (Participants) | 42 | 42 | 42
percentage of participants | 38.1 | 31.0 | 35.7

11. Secondary Outcome: Percentage of Study Participants With Serious Treatment-emergent Adverse Events (TEAEs) in Part A
Description: as for outcome 5
Time Frame: From Baseline (Day 1) to Safety Follow-up Period of Part A (up to Day 39)
Population: SS A included all study participants who were randomized and received full or partial study medication according to the treatment that the participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: UCB0599: Capsule 180 mg | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599: Encapsulated Tablet 180 mg
Number analyzed (Participants) | 42 | 42 | 42
percentage of participants | 0 | 0 | 0

12. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From Study in Part A
Time Frame: From Baseline (Day 1) to Safety Follow-up Period of Part A (up to Day 39)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Part A: UCB0599: Capsule 180 mg | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599: Encapsulated Tablet 180 mg
Number analyzed (Participants) | 42 | 42 | 42
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For Part A: From Baseline (Day 1) of Part A until Safety Follow-Up (up to Day 39) and for Part B: From Baseline (Day 1) to Safety Follow-up Period of Part B (up to Day 15)
Description: Treatment emergent AEs (TEAE): all AEs starting on/after the date/time of first treatment & up to including 4 days after last treatment or any unresolved event already present before administration of treatment that worsens in intensity following exposure to treatment. Safety Sets (Part A & B) included All study participants who were randomized and received full or partial study medication according to the treatment that the participants actually received.
Groups:
- Part A: UCB0599 180 mg/Day Capsules: All participants who received a single dose of UCB0599 180 mg capsule under fasting conditions on Day 1 in Period 1 (normal gastric pH), Day 19 in Period 4 (elevated gastric pH), Day 11 in Period 3 (normal gastric pH), Day 29 in Period 6 (elevated gastric pH), Day 6 in Period 2 (normal gastric pH), and Day 24 in Period 5 (elevated gastric pH). Esomeprazole was coadministered with UCB0599 180 mg capsule in Treatment Periods 4, 5, and 6 (elevated gastric pH).
- Part A: UCB0599 180 mg/Day Encapsulated Tablets: All participants who received a single dose of UCB0599 180 mg encapsulated tablet under fasting conditions on Day 1 in Period 1 (normal gastric pH), Day 19 in Period 4 (elevated gastric pH), Day 6 in Period 2 (normal gastric pH), Day 24 in Period 5 (elevated gastric pH), Day 11 in Period 3 (normal gastric pH), and Day 29 in Period 6 (elevated gastric pH). Esomeprazole was coadministered with UCB0599 180 mg encapsulated tablet in Treatment Periods 4, 5, and 6 (elevated gastric pH).
- Part B: UCB0599 360mg (Japanese Participants): Japanese participants who received a single dose of UCB0599 360 mg capsule on Day 1 of Period 1 and Day 6 of Period 2. Period 1 and Period 2 were separated by a washout period of 4 days.
Arm/Group | Part A: UCB0599 180 mg/Day Capsules | Part A: UCB0599: Non-encapsulated Tablet 180 mg | Part A: UCB0599 180 mg/Day Encapsulated Tablets | Part B: Pooled Placebo (Japanese Participants) | Part B: UCB0599 90 mg (Japanese Participants) | Part B: UCB0599 180 mg (Japanese Participants) | Part B: UCB0599 360mg (Japanese Participants) | Part B: Pooled Placebo (Chinese Participants) | Part B: UCB0599 90 mg (Chinese Participants) | Part B: UCB0599 180 mg (Chinese Participants) | Part B: UCB0599 360 mg (Chinese Participants)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/42 | 0/3 | 0/8 | 0/8 | 0/8 | 0/3 | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42 | 0/3 | 0/8 | 0/8 | 0/8 | 0/3 | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 5/42 | 11/42 | 6/42 | 1/3 | 2/8 | 0/8 | 0/8 | 1/3 | 1/8 | 3/9 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: UCB0599 180 mg/Day Capsules (N=42) | Part A: UCB0599: Non-encapsulated Tablet 180 mg (N=42) | Part A: UCB0599 180 mg/Day Encapsulated Tablets (N=42) | Part B: Pooled Placebo (Japanese Participants) (N=3) | Part B: UCB0599 90 mg (Japanese Participants) (N=8) | Part B: UCB0599 180 mg (Japanese Participants) (N=8) | Part B: UCB0599 360mg (Japanese Participants) (N=8) | Part B: Pooled Placebo (Chinese Participants) (N=3) | Part B: UCB0599 90 mg (Chinese Participants) (N=8) | Part B: UCB0599 180 mg (Chinese Participants) (N=9) | Part B: UCB0599 360 mg (Chinese Participants) (N=8)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 7 (7) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT05845645/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT05845645/SAP_001.pdf